CLINICAL TRIAL: NCT06500611
Title: Combined Effects Of Sensory Integration And Vestibular Exercises On Dizziness, Fall Risk And Quality Of Life In Post-Stroke Patients
Brief Title: Combined Effects Of Sensory Integration And Vestibular Exercises On Post-Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0271
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Post Stroke
Keywords: sensory integration,; stroke; vestibular rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Sensory Integration and Vestibular Exercise with Routine Physical Therapy) (Experimental): Sensory Integration Exercise:
  Week 1-2
  1. Eyes Open Standing for 5 minutes.
  2. Sitting position for 5 minutes.
  Week 3-4
  1. Eyes Closed Standing for 5 minutes.
  2. Sit to stand for 5 minutes.
  Week 5-6
  1. Tandem Walk for 4 minutes.
  2. Walk Obstacle Course for 4 minutes.
  Vestibular Exercise
  Week 1-2
  1. Head Movements for 5 minutes
  2. Gaze Stabilization for 5 minutes.
  Week 3-4
  1. Single Leg Stance for 5 minutes.
  2. Rotation Exercises for 5 minutes.
  Week 5-6
  1. Walking Patterns for 4 minutes.
  2. Pendulum Exercise for 4 minutes.
  3. Catch and Throw for 4 minutes.
  Routine Physical Therapy for 20 minutes.
  Interventions: Other: Sensory Integration and Vestibular Exercise with Routine Physical Therapy
- GROUP B (Vestibular Exercise with Routine Physical Therapy) (Experimental): Vestibular Exercise
  Week 1-2
  1. Head Movements for 10 minutes
  2. Gaze Stabilization for 10 minutes.
  Week 3-4
  1. Single Leg Stance for 10 minutes.
  2. Rotation Exercises for 10 minutes.
  Week 5-6
  1. Walking Patterns for 5 minutes.
  2. Pendulum Exercise for 5 minutes.
  3. Catch and Throw for 10 minutes.
  Routine Physical Therapy for 20 minutes.
  Interventions: Other: Vestibular Exercise with Routine Physical Therapy

INTERVENTIONS:
Other: Sensory Integration and Vestibular Exercise with Routine Physical Therapy — 1. Stand with feet hip-width apart 5 rep
  2. Sit in chair without backrest 5 rep
  1.Stand with feet hip -width apart 5 rep
  2.Sit to stand sit on chair without backrest and perform sit to stand repeatedly 5 rep
  1.Tandem Walk one foot directly in front of the other.2 sets 5 steps forward and backward
  2.Patientwalk forward cross an obstacle, continue walk. Walk Lateral Walk Backward 2 sets
  1. Stand and slowly move head side to side and up down 10 repetition
  2. Fix gaze and move head side to side or up and down 10 repetitions
  1. Stand on one leg for 10 seconds hold on. Repeat 5 times on each leg.
  2. Stand and rotate body to right and left 10 rotations
  1. Walk on straight line , zigzag pattern, walk while looking your shoulder 5 rep
  2. Sit and swing your legs back and forth 5rep
  3. Play catch in standing. 2 sets 5-8 catches.
  Static stretching 30 sec hold 5 times
  Arms: GROUP A (Sensory Integration and Vestibular Exercise with Routine Physical Therapy)
Other: Vestibular Exercise with Routine Physical Therapy — Vestibular exercise
  1. Stand with feet hip -width apart and slowly move head side to side and up down.10 repetitions for each direction.
  2 .Fix your gaze on object while moving your head side to side or up and down. 10 repetitions for each movement.
  1.Patient will stand on one leg for 10 second. Hold onto a stable support if needed. 5 times on each leg.
  2. Stand with feet hip-width apart and rotate body to the right and left. 10 rotations in each direction.
  1. Walk on a straight line or in a zigzag pattern or walk while looking over your shoulder. (5 rep)
  2. Sit on a stable chair and swing your legs back and forth, similar to a pendulum. (5rep)
  3. Catch and Throw play catch with a partner while standing. 2 sets of 5-8 catches.
  Routine Physical Therapu Static stretching exercises for 30 sec hold with 30 sec rest. 5 times for each muscle group
  Arms: GROUP B (Vestibular Exercise with Routine Physical Therapy)

SUMMARY:
The aim of this study is to determine the combined effects of sensory integration and vestibular exercise on dizziness, fall risk and quality of life.

DETAILED DESCRIPTION:
This randomized controlled trial will be conducted at Mansoorah Teaching Hospital in 7 months after the approval of the synopsis. 38 participants with stroke will be included as per the sample size calculation through the convenience sampling technique. Participants who meet inclusion criteria will be randomly allocated using an online randomization tool into two groups Group A will receive Combine Sensory integration exercise and vestibular exercise with routine physical therapy for 40 minutes and Group B will receive Vestibular exercise with routine physical therapy for 40 minutes. Each group will receive a treatment session of 3 times in week for 6 weeks. The data will be analyzed using SPSS version 24.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age between 40years-65years
* those who have been diagnosed with vestibular disorders
* An ability to stand for for 5 minutes without aid measured by 5 times sit to stand test.

Exclusion Criteria:

* Have bilateral or unstable vestibular loss
* Any neurological condition is present
* Active BPPV is present
* Any acute orthopaedic condition is present
* Peripheral neuropathy is present
* Visual impairment not corrected with glasses.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Combined Effects Of Sensory Integration And Vestibular Exercises On Post-Stroke Patients | 6 weeks
  DHI assesses Dizziness Consists 25 items three answers yes sometimes no. Highest disability 100 ,lowest one be 0.The SS-QOL, disease-specific consist 49 items 12 domains, social role (five questions), mobility (six questions), energy (three questions), language (five questions), self-care (five questions), mood (five questions), personality (three questions), thinking (three questions), upper extremity function (five questions), family role (three questions), vision (three questions),work/productivity (three questions). Each item ranked five-point level one means completely agreed while level five means completely disagree. Total score ranges from 49 to 245.Time up and go test Duration of ≥13.5 s associate increased fall risk with vestibular dysfunction. STRATIFY tool comprises five items risk factors past history falling, patient agitation, visual impairment, incontinence, transfer and mobility score range from 0 to 5 points and risk of falling is a score ≥ 2 points.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehab Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He A, Wang Z, Wu X, Sun W, Yang K, Feng W, Wang Y, Song H. Incidence of post-stroke cognitive impairment in patients with first-ever ischemic stroke: a multicenter cross-sectional study in China. Lancet Reg Health West Pac. 2023 Jan 14;33:100687. doi: 10.1016/j.lanwpc.2023.100687. eCollection 2023 Apr. PMID 37181529
- [Background] Harjpal P, Qureshi MI, Kovela RK, Jain M. Efficacy of Bilateral Lower-Limb Training Over Unilateral Lower-Limb Training To Reeducate Balance and Walking in Post-Stroke Survivors: A Randomized Clinical Trial. Cureus. 2022 Oct 27;14(10):e30748. doi: 10.7759/cureus.30748. eCollection 2022 Oct. PMID 36447690
- [Background] Einstad MS, Saltvedt I, Lydersen S, Ursin MH, Munthe-Kaas R, Ihle-Hansen H, Knapskog AB, Askim T, Beyer MK, Naess H, Seljeseth YM, Ellekjaer H, Thingstad P. Associations between post-stroke motor and cognitive function: a cross-sectional study. BMC Geriatr. 2021 Feb 5;21(1):103. doi: 10.1186/s12877-021-02055-7. PMID 33546620
- [Background] Zhou Z, Lu J, Liu WW, Manaenko A, Hou X, Mei Q, Huang JL, Tang J, Zhang JH, Yao H, Hu Q. Advances in stroke pharmacology. Pharmacol Ther. 2018 Nov;191:23-42. doi: 10.1016/j.pharmthera.2018.05.012. Epub 2018 May 25. PMID 29807056
- [Background] Rodriguez-Fernandez A, Lobo-Prat J, Font-Llagunes JM. Systematic review on wearable lower-limb exoskeletons for gait training in neuromuscular impairments. J Neuroeng Rehabil. 2021 Feb 1;18(1):22. doi: 10.1186/s12984-021-00815-5. PMID 33526065
- [Background] Li S, Francisco GE, Zhou P. Post-stroke Hemiplegic Gait: New Perspective and Insights. Front Physiol. 2018 Aug 2;9:1021. doi: 10.3389/fphys.2018.01021. eCollection 2018. PMID 30127749
- [Background] Rodgers H, Bosomworth H, Krebs HI, van Wijck F, Howel D, Wilson N, Finch T, Alvarado N, Ternent L, Fernandez-Garcia C, Aird L, Andole S, Cohen DL, Dawson J, Ford GA, Francis R, Hogg S, Hughes N, Price CI, Turner DL, Vale L, Wilkes S, Shaw L. Robot-assisted training compared with an enhanced upper limb therapy programme and with usual care for upper limb functional limitation after stroke: the RATULS three-group RCT. Health Technol Assess. 2020 Oct;24(54):1-232. doi: 10.3310/hta24540. PMID 33140719
- [Background] Brown KE, Neva JL, Feldman SJ, Staines WR, Boyd LA. Sensorimotor integration in chronic stroke: Baseline differences and response to sensory training. Restor Neurol Neurosci. 2018;36(2):245-259. doi: 10.3233/RNN-170790. PMID 29526859
- [Background] Krishnan K, Bassilious K, Eriksen E, Bath PM, Sprigg N, Braekken SK, Ihle-Hansen H, Horn MA, Sandset EC. Posterior circulation stroke diagnosis using HINTS in patients presenting with acute vestibular syndrome: A systematic review. Eur Stroke J. 2019 Sep;4(3):233-239. doi: 10.1177/2396987319843701. Epub 2019 Apr 10. PMID 31984230
- [Background] Regauer V, Seckler E, Muller M, Bauer P. Physical therapy interventions for older people with vertigo, dizziness and balance disorders addressing mobility and participation: a systematic review. BMC Geriatr. 2020 Nov 23;20(1):494. doi: 10.1186/s12877-020-01899-9. PMID 33228601
- [Background] Lubetzky AV, Kelly J, Wang Z, Gospodarek M, Fu G, Sutera J, Hujsak BD. Contextual sensory integration training via head mounted display for individuals with vestibular disorders: a feasibility study. Disabil Rehabil Assist Technol. 2022 Jan;17(1):74-84. doi: 10.1080/17483107.2020.1765419. Epub 2020 May 18. PMID 32421374
- [Background] Ekvall Hansson E, Pessah-Rasmussen H, Bring A, Vahlberg B, Persson L. Vestibular rehabilitation for persons with stroke and concomitant dizziness-a pilot study. Pilot Feasibility Stud. 2020 Sep 30;6:146. doi: 10.1186/s40814-020-00690-2. eCollection 2020. PMID 33005434
- [Background] Xie G, Wang T, Jiang B, Su Y, Tang X, Guo Y, Liao J. Effects of hydrokinesitherapy on balance and walking ability in stroke survivors: a systematic review and meta-analysis of randomized controlled studies. Eur Rev Aging Phys Act. 2019 Nov 13;16:21. doi: 10.1186/s11556-019-0227-0. eCollection 2019. PMID 31754406
- [Background] Meng L, Liang Q, Yuan J, Li S, Ge Y, Yang J, Tsang RCC, Wei Q. Vestibular rehabilitation therapy on balance and gait in patients after stroke: a systematic review and meta-analysis. BMC Med. 2023 Aug 25;21(1):322. doi: 10.1186/s12916-023-03029-9. PMID 37626339
- [Background] Lubetzky AV, Harel D, Krishnamoorthy S, Fu G, Morris B, Medlin A, Wang Z, Perlin K, Roginska A, Cosetti M, Kelly J. Decrease in head sway as a measure of sensory integration following vestibular rehabilitation: A randomized controlled trial. J Vestib Res. 2023;33(3):213-226. doi: 10.3233/VES-220107. PMID 36911951
- [Background] Ghaffari A, Asadi B, Zareian A, Akbarfahimi M, Raissi GR, Fathali Lavasani F. The Effects of Vestibular Rehabilitation on Poststroke Fatigue: A Randomized Controlled Trial Study. Stroke Res Treat. 2022 Aug 31;2022:3155437. doi: 10.1155/2022/3155437. eCollection 2022. PMID 36090743
- [Background] Tramontano M, Russo V, Spitoni GF, Ciancarelli I, Paolucci S, Manzari L, Morone G. Efficacy of Vestibular Rehabilitation in Patients With Neurologic Disorders: A Systematic Review. Arch Phys Med Rehabil. 2021 Jul;102(7):1379-1389. doi: 10.1016/j.apmr.2020.11.017. Epub 2020 Dec 28. PMID 33383031
- [Background] Mitsutake T, Imura T, Tanaka R. The Effects of Vestibular Rehabilitation on Gait Performance in Patients with Stroke: A Systematic Review of Randomized Controlled Trials. J Stroke Cerebrovasc Dis. 2020 Nov;29(11):105214. doi: 10.1016/j.jstrokecerebrovasdis.2020.105214. Epub 2020 Aug 8. PMID 33066892
- [Background] Gandolfi M, Vale N, Dimitrova E, Zanolin ME, Mattiuz N, Battistuzzi E, Beccari M, Geroin C, Picelli A, Waldner A, Smania N. Robot-Assisted Stair Climbing Training on Postural Control and Sensory Integration Processes in Chronic Post-stroke Patients: A Randomized Controlled Clinical Trial. Front Neurosci. 2019 Oct 24;13:1143. doi: 10.3389/fnins.2019.01143. eCollection 2019. PMID 31708735
- [Background] Adomaviciene A, Daunoraviciene K, Kubilius R, Varzaityte L, Raistenskis J. Influence of New Technologies on Post-Stroke Rehabilitation: A Comparison of Armeo Spring to the Kinect System. Medicina (Kaunas). 2019 Apr 9;55(4):98. doi: 10.3390/medicina55040098. PMID 30970655
- [Background] Kelly J, Harel D, Krishnamoorthy S, Fu G, Morris B, Medlin A, Mischinati S, Wang Z, Sutera J, Perlin K, Cosetti M, Lubetzky AV. Contextual sensory integration training vs. traditional vestibular rehabilitation: a pilot randomized controlled trial. J Neuroeng Rehabil. 2023 Aug 12;20(1):104. doi: 10.1186/s12984-023-01224-6. PMID 37568216
- [Background] Jang SH, Lee JH. Impact of sensory integration training on balance among stroke patients: sensory integration training on balance among stroke patients. Open Med (Wars). 2016 Aug 13;11(1):330-335. doi: 10.1515/med-2016-0061. eCollection 2016. PMID 28352817
- [Background] Tamber AL, Wilhelmsen KT, Strand LI. Measurement properties of the Dizziness Handicap Inventory by cross-sectional and longitudinal designs. Health Qual Life Outcomes. 2009 Dec 21;7:101. doi: 10.1186/1477-7525-7-101. PMID 20025754
- [Background] Mahmoodi M, Safari A, Vossoughi M, Golbon-Haghighi F, Kamali-Sarvestani M, Ghaem H, Borhani-Haghighi A. Stroke specific quality of life questionnaire: Test of reliability and validity of the Persian version. Iran J Neurol. 2015 Apr 4;14(2):94-100. PMID 26056554
- [Background] Alghadir AH, Al-Eisa ES, Anwer S, Sarkar B. Reliability, validity, and responsiveness of three scales for measuring balance in patients with chronic stroke. BMC Neurol. 2018 Sep 13;18(1):141. doi: 10.1186/s12883-018-1146-9. PMID 30213258
- [Background] Aranda-Gallardo M, Enriquez de Luna-Rodriguez M, Vazquez-Blanco MJ, Canca-Sanchez JC, Moya-Suarez AB, Morales-Asencio JM. Diagnostic validity of the STRATIFY and Downton instruments for evaluating the risk of falls by hospitalised acute-care patients: a multicentre longitudinal study. BMC Health Serv Res. 2017 Apr 17;17(1):277. doi: 10.1186/s12913-017-2214-3. PMID 28412939
- [Background] Choi JU, Kang SH. The effects of patient-centered task-oriented training on balance activities of daily living and self-efficacy following stroke. J Phys Ther Sci. 2015 Sep;27(9):2985-8. doi: 10.1589/jpts.27.2985. Epub 2015 Sep 30. PMID 26504340
- [Background] Ricci NA, Aratani MC, Caovilla HH, Gananca FF. Effects of Vestibular Rehabilitation on Balance Control in Older People with Chronic Dizziness: A Randomized Clinical Trial. Am J Phys Med Rehabil. 2016 Apr;95(4):256-69. doi: 10.1097/PHM.0000000000000370. PMID 26368833